CLINICAL TRIAL: NCT00289003
Title: An Exploratory, Randomised, Parallel Group Study, Comparing the Protective Effect of Soluble Beta-1,3/1,6-Glucan or Placebo in Oral Mucositis in Head and Neck Cancer Patients Receiving Radiation Therapy or Chemoradiotherapy
Brief Title: The Protective Effect of Soluble Beta-1,3/1,6-Glucan Compared to Placebo in Oral Mucositis in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMR-907-SBG-1-02-HN
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2006-05

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

INTERVENTIONS:
Drug: Soluble beta-1,3/1,6-glucan

SUMMARY:
The purpose of this study is to explore the protective effect and safety of soluble beta-1,3/1,6-glucan compared to placebo in oral mucositis in head and neck patients receiving radiotherapy or chemoradiotherapy.

Hypothesis: Soluble beta-1,3/1,6-glucan will through its immunomodulating activities prevent oral mucositis

DETAILED DESCRIPTION:
Oral mucositis is defined as inflammation and ulceration of the mucous membranes of the mouth. The condition is very painful and might put the patient at risk of serious systemic infections and is a common dose-limiting toxicity of chemotherapy and radiotherapy. The present treatment of mucositis is primarily supportive; strong analgesics in addition to oral hygiene. Prophylactic antibiotics have been used and many topical agents are available to palliate mucositis, but no standard therapy has been accepted.

Comparison: Methyl cellulose has been chosen as placebo due to its close resemblance to soluble beta-1,3/1,6-glucan in terms of general appearance and viscosity. Methyl cellulose is a viscous solution which might form a mucosal barrier. Physical barriers are considered having a protective function in oral mucositis, and methyl cellulose might be considered as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiotherapy or chemoradiotherapy for histologically confirmed squamous cell carcinoma of oral cavity or oropharynx (1.8-2.0 Gy/day; 5 days per week, totally 59.4-70 Gy).
* Normal mucosa at baseline (i.e. Common Toxicity Criteria (CTC) grade 0)
* >= 18 years of age
* Women of childbearing potential must use an adequate contraceptive method and have a negative pregnancy test
* Written informed consent

Exclusion Criteria:

* Patients who will receive hyperfractionated or accelerated radiotherapy
* History of malignancies within the past five years other than non-melanomatous skin cancers (with the exception of squamous cell carcinoma of the skin) or carcinoma in situ of the cervix
* Previous neoplasm in the head and neck area, whether malignant or not
* Previous radiation therapy for head and neck cancer
* If wound from curative surgery have not healed
* Patients expected to receive agents that would interfere with the investigator's ability to assess changes in the appearance of the mucositis during the study
* Use of radiosensitizers
* History or clinical evidence of active significant acute or chronic diseases that may compromise the ability to evaluate or interpret the effects of the study treatment on mucositis
* Evidence of distant metastatic disease
* Expected survival of less than 12 months
* > grade 3 performance status (WHO grading)
* Granulocyte count < 2.000/mm3 and platelet count < 100,000/mm3
* Serum creatinine >= 150 micromol/L
* Total bilirubin >= 36 micromol/L, AST > 3 times the upper normal limit
* Any subject who, in the opinion of the investigator, is unlikely to comply with the study procedures, or is unlikely to complete the study due to different reasons like e.g. language barriers or mental incapacity
* Participation in a clinical trial in the last 30 days Receipt of any investigational product within 30 days prior to this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-10; Study Completion 2006-07

PRIMARY OUTCOMES:
To assess actual grade of mucositis upon completion of radiotherapy or chemoradiotherapy and after prophylactic treatment with soluble beta-1,3/1,6-glucan or placebo.

SECONDARY OUTCOMES:
To assess proportions of patients avoiding grade 2 or higher oral mucositis after treatment with soluble beta-1,3/1,6-glucan or placebo
To assess time before first sign of oral mucositis
To evaluate impact of toxicities like patients' pain and swallowing difficulty
To assess the safety of the investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Nutting, Dr.med., Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (3):
- Germany (2):
  - Medical Centre Bonn, Clinic for Radiotherapy and Radiological Oncology, Bonn
  - Evangelisches Krankenhaus, Düsseldorf
- Royal Marsden Hospital, Head and Neck Unit, London, United Kingdom